CLINICAL TRIAL: NCT04075851
Title: The Prevalence of Serum Thyroid Hormone Autoantibodies in Autoimmune Thyroid Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Hai-qing Zhang, Professor, Shandong Provincial Hospital
Other Study IDs: 20190801
Record Dates: First submitted 2019-08-29; First posted 2019-09-03 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Autoimmune Thyroid Disease
Keywords: Autoimmune thyroid disease; Thyroid hormone autoantibodies; Hashimoto's thyroiditis; Grave's disease
MeSH Terms: conditions — Hashimoto Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Hashimoto or Grave's disease patients in treatment: Draw 10 ml venous blood
- Hashimoto or Grave's disease patients on initial treatment: 10 ml of venous blood was extracted every month for three months
- Pregnant woman with Hashimoto or Grave's disease: 10 ml venous blood was extracted every month to postpartum for 6 months
- Healthy crowd: Draw 10 ml venous blood

SUMMARY:
Thyroid hormone autoantibodies(THAA) in serum can Interfere radioimmunoassay for the determination of free thyroid hormones. Thyroid function test plays a key role in the diagnosis and treatment of autoimmune thyroid disease (AITD), and abnormal examination results in misdiagnosis and mistreatment. At present, the epidemiological results of THAA in AITD are inconsistent, and the pathogenesis has not been clarified. However, there is no relevant research on THAA in China. This project intends to collect AITD patients and healthy people, detecting THAA, at the same time testing thyroid function and thyroid autoantibodies, definiting positive rate of THAA in AITD patients, observing the effect of common therapeutic drugs for AITD on THAA, investigating the rule of THAA influencing thyroid function test results .This project will provide the basis and method for how to effectively avoid THAA interfering with thyroid function test.

ELIGIBILITY:
Inclusion Criteria:

* male or female with Hashimoto thyroiditis or Grave's disease aged for 18 to 65 years old

Exclusion Criteria:

* Had a thyroidectomy Had a thyroid fine needle puncture biopsy Autoimmune diseases Take drugs that affect the immune system

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Autoimmune thyroid diseases in endocrine outpatient department of shandong provincial hospital from August 1, 2019 to August 1, 2022
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
prevalence of thyroid hormone autoantibodies in AITD | measured after 1 year of follow-up
  Radioimmuno precipitation test used for thyroid hormone autoantibodies

CONTACTS AND LOCATIONS:
Overall Officials: Haiqing Zhang, Study Chair — shandong province hospital
Locations (1):
- Shandong Province Hospital, Jinan, Shandong, China